CLINICAL TRIAL: NCT02866084
Title: Neuromodulation Treatment of Vestibular Migraines
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Scion NeuroStim (Industry)
Responsible Party: Principal Investigator, Michael E. Hoffer, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160566
Record Dates: First submitted 2016-08-05; First posted 2016-08-15 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Headache
Keywords: vestibular migraines; dizziness; migraine headache
MeSH Terms: conditions — Headache; Dizziness; Migraine Disorders | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device (Experimental): Neuromodulation
  Interventions: Device: Device

INTERVENTIONS:
Device: Device — The following parameters will be set for active treatments using the CVS Device:
  * A standardized CVS time-varying waveform lasting approximately 19 minutes will be used. Treatments will be administered up to twice daily. The two daily treatments should ideally be separated by at least one hour.
  * The waveform schedule will consist of a warm sawtooth delivered to one ear and a cold sawtooth delivered to the other ear. The warm sawtooth will go from body temperature to 42 °C, and the cold sawtooth will go from body temperature to 17 °C. The two waveforms will be delivered simultaneously, but will have different oscillation frequencies.
  Other Names: Caloric stimulation

SUMMARY:
This is a non-randomized pilot study to test the efficacy of neuromodulation via caloric stimulation on vestibular migraines. All subject who meet the study criteria will be in an active treatment group. All subjects will report the frequency of the migraines and undergo periodic testing of symptoms.

DETAILED DESCRIPTION:
This is a non-blinded, non-randomized pilot study of individuals with vestibular migraines. The goal is to test the efficacy of neuromodulation on both migraine and dizziness symptoms in patients with documented vestibular migraines. Treatment will consist of 9 months of active treatment followed by 3 months of observation. The active treatment requires two daily 20 minute sessions wearing a device over the ears that delivers a very small amount of warm air to the ears. All subjects will undergo a series of tests at baseline and at discrete intervals during the 1 year of observation.

Primary and Secondary endpoints are listed below:• Primary Efficacy Endpoints

1. Reduction in the frequency and severity of migraine headaches (self reported in pain diary)
2. Reduction in the frequency and intensity of perceived vestibular symptoms (Dizziness Handicap Inventory (DHI), Activity Balance confidence scale (ABC), Oscillopsia Test, Symptoms questionnaire), OVRT Goggle profile.

Secondary Efficacy Endpoints for the Pilot Study

1. Improvement in sleep quality and/or quantity as assessed by the Epworth Sleep Scale.
2. Improvement in quality of life as assessed by the HIT-6 survey.
3. Improvement in mood/anxiety as assessed with the T2 Mood Tracker app (National Center for Telehealth & Technology).

ELIGIBILITY:
Inclusion Criteria:

1. Adults, between the ages of 18 and 75 who have been diagnosed with VM least 3 months prior to entering into the study.
2. The Investigator must have confidence in the patient's ability to reliably use the CVS Device and complete the requirements of the study.

Exclusion Criteria:

1. are pregnant
2. have a history of cardiovascular disease
3. work night shifts
4. have a history of unstable mood disorder or unstable anxiety disorder
5. use a hearing aid
6. have a cochlear implant
7. abuse alcohol or other drugs
8. are experiencing Medication Overuse Headaches (individuals with respect to whom the Investigator is concerned that analgesic abuse is involved based on the ICHD-II guidelines).
9. have had eye surgery within the previous three months or ear surgery within the previous six months
10. have active ear infections or a perforated tympanic membrane
11. have participated in another clinical trial within the last 30 days or are currently enrolled in another clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory | Until study completion up to 12 months
  Questionnaire of dizziness symptoms
Headache Impact Test | Until study completion up to 12 months
  Headache questionnaire
Activities Balance Confidence Interval | Until study completion up to 12 months
  Dizziness questionnaire
OVRT Testing | Until study completion up to 12 months
  Oculomotor, vestibular, and reaction time tests

SECONDARY OUTCOMES:
Epworth Sleepiness Scale | Until study completion up to 12 months
  Sleepiness questionnaire
T2 Mood Tracker app | Until study completion up to 12 months
  App to assess mood and anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saper JR, Dodick DW, Silberstein SD, McCarville S, Sun M, Goadsby PJ; ONSTIM Investigators. Occipital nerve stimulation for the treatment of intractable chronic migraine headache: ONSTIM feasibility study. Cephalalgia. 2011 Feb;31(3):271-85. doi: 10.1177/0333102410381142. Epub 2010 Sep 22. PMID 20861241
- [Background] Tedeschi G, Russo A, Conte F, Laura M, Tessitore A. Vestibular migraine pathophysiology: insights from structural and functional neuroimaging. Neurol Sci. 2015 May;36 Suppl 1:37-40. doi: 10.1007/s10072-015-2161-x. PMID 26017509